CLINICAL TRIAL: NCT04685161
Title: Comparison of Surgical Extrusion vs Fibre Post Restoration for Crown-root Fractured Maxillary Incisors. Randomized Clinical Trial
Brief Title: Comparison of Surgical Extrusion vs. Fibre Post Restoration for Crown-root Fractured Maxillary Incisors.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tamil Nadu Dr.M.G.R.Medical University (Other)
Responsible Party: Principal Investigator, Rahul Baskar, Principal investigator, Tamil Nadu Dr.M.G.R.Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSICOLLEGE
Record Dates: First submitted 2020-12-16; First posted 2020-12-28 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Fractured Tooth
MeSH Terms: conditions — Tooth Fractures

STUDY DESIGN:
Intervention Model Description: 2 groups are used One using fibre post placement And the other using surgical extrusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical extrusion (Experimental): Novel and alternative treatment option for horizontal crown root fractured maxillary incisors
  Interventions: Procedure: Surgical extrusion
- Fibre post (Active Comparator): Treatment modality normally used for crown-root fractured tooth
  Interventions: Device: Fibre post

INTERVENTIONS:
Procedure: Surgical extrusion — Invasive treatment option for fractured tooth
  Arms: Surgical extrusion
Device: Fibre post — Easy approach for treatment
  Arms: Fibre post

SUMMARY:
A total of 124 samples was calculated to be sufficient with G*power software ver 3.1.9.2 with effect size of 0.4 alpha probability error and power 0.95.With drop out estimate of 10% the final sample size decided was 140 samples. Patients reporting with complicated(pulp exposed or pulpally involved) horizontal crown root fracture with loss of crown structure in maxillary incisors and radiograph evidence of supra alveolar tooth structure are recruited for study. Informed consent from the patients or guardian as appropriate is obtained as suitable prior to treatment delivery. Exclusion criteria were:patients not willing for recall visits, root with evidence of cervical resorption or roor canal filling, open apices, patient with systemic ailments rendering root canal treatment, compromised periodontal health, vertical or horizontal root fracture. Pulpal condition of tooth was assessed using cold sensibility test(Neosnow, orikam health care Ltd, India.) amd confirmed upon access opening with teeth showing evidence of pulpal bleeding wad categorized as irreversible pulpitis and teeth with no evidence of pulpal bleeding categorized as necrotic pulp.

DETAILED DESCRIPTION:
Patients are randomly alloted to treatment groups. Group I-Root canal treatment followed by surgical extrusion of teeth till about 40%supra gingival crown structure is visible clinically.

Group II-Root canal treatment followed by glass fibre post placement (Reforpost, Angelus, Brazil) and composite (charisma smart, Germany) core build up with porcelain fused metal crown.

Post treatment visits are scheduled 6,12,18 months, scheduled visits were planned as close as possible to the study protocol, but for the purpose of data collection, any recall visit occuring within plus or minus 10% of the advocated time was considered aa occuring at that time. Recall visit check up included clinical examination for mobility, periapical tenderness, gingival pocket depth estimation,bleeding on probing and radiographic examination. Patients are asked to report immediately of any unforeseen circumstances arises in the restored teeth.

ELIGIBILITY:
Inclusion Criteria:

* patients with complicated crown root fracture
* patients willing for recall
* Good oral hygiene

Exclusion Criteria:

* patients not willing for recall
* Patients health rendering root canal treatment

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Radiographic healing of teeth is measured | 18 months
  Periapical index score(PAI) is used for assessment

CONTACTS AND LOCATIONS:
Overall Officials: ANAND SHERWOOD, MDS, Study Director — TNMGRMU
Locations (1):
- Csi College of Dental Sciences and Research, Madurai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No